CLINICAL TRIAL: NCT05177185
Title: A Phase 2 Prospective Trial of Hippocampal-Sparing Stereotactic Radiosurgery Treatment of Brain Metastases Using CyberKnife
Brief Title: Hippocampal-Sparing Stereotactic Radiosurgery Treatment of Brain Metastases Using CyberKnife
Acronym: HiSparCK
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200253-01H
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Brain Metastases; Radiosurgery
Keywords: Hippocampal-sparing
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: All patients will undergo hippocampal-sparing stereotactic radiosurgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SRS with hippocampal-sparing (Experimental): Stereotactic radiosurgery with hippocampal-sparing
  Interventions: Radiation: Hippocampal-sparing; Radiation: Stereotactic radiosurgery

INTERVENTIONS:
Radiation: Hippocampal-sparing — Dose constraint placed on hippocampi to minimize dose to hippocampi, while maintaining target coverage (at least 98% of brain metastasis volume must receive 100% of prescription dose).
Radiation: Stereotactic radiosurgery — Stereotactic radiosurgery (SRS) with prescription dose determined based on size of brain metastasis; 21 or 24 Gy in a single fraction if less than or equal to 20 mm, 18Gy in a single fraction in 21 - 30 mm, 15 Gy in a single fraction or 30 Gy in 5 fractions if 31 - 40 mm (physician discretion).
  Other Names: SRS; Stereotactic radiotherapy

SUMMARY:
This phase II clinical trial involves the use of hippocampal-sparing together with stereotactic radiosurgery (SRS) for the treatment of brain metastases. The standard of care in the treatment of brain metastases is cranial radiation, but this can be associated with significant neurocognitive sequelae, including reduced verbal memory, spatial memory, attention and problem solving. This can be minimized with the use of SRS, rather than whole brain radiotherapy (WBRT).

Additionally, some of the neurotoxicity has been linked to damage in neural progenitor cells contained within the hippocampus. A recent phase III clinical trial has demonstrated reduced neurocognitive decline with use of hippocampal-sparing techniques in WBRT. This trial aims to see if this can be further improved by combining SRS and hippocampal-sparing.

DETAILED DESCRIPTION:
Primary objective: To determine the rate of neurocognitive failure with hippocampal-sparing stereotactic radiosurgery compared to neurocognitive failures rates with hippocampal-sparing whole brain radiotherapy (using NRG-CC001 with the same population as our comparison), assessed at baseline and at months 3, 6 and 12 (+/- 2 weeks), and with failure defined as any decline in at least one of the following tests (of note, we will be using alternate forms to avoid practice effects): Hopkins Verbal Learning Test for total recall, delayed recall and delayed recognition, Controlled oral word association, Trail making tests parts A and B, Brief visuospatial memory test-revised.

Secondary objectives:

(I) To determine if hippocampal-sparing preserves neurocognitive function, assessed at baseline and months 3, 6 and 12 (+/- 2 weeks), and defined as decline in at least one of the following tests (of note, we will be using alternate forms to avoid practice effects): Hopkins Verbal Learning Test for total recall, delayed recall and delayed recognition, Controlled oral word association, Trail making tests parts A and B, Brief visuospatial memory test-revised.

(II) To determine the incidence of adverse events up to 12 months post-treatment, as measured by common terminology criteria for adverse events (CTCAE v3.0) (III) Quality of life As measured using MD Anderson Symptom Inventory for Brain tumor (MDASI-BT)'s four subscales: symptom severity, symptom interference, neurologic failure and cognitive factor score; and individual items (fatigue, neurologic factor items and cognitive factor items).

(III) Oncologic outcomes will also be assessed at surveillance every 3 months, as is standard of care; time to intracranial progression, overall survival. These will be estimated using Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Either gender
* Patients must provide informed consent prior to registration
* Pathologically (histologically or cytologically) proven diagnosis of solid tumor malignancy
* Brain metastase(s) outside a 5-mm margin around either hippocampus
* Brain metastase(s) must be visible on contrast-enhanced magnetic resonance imaging (MRI); an allowed exception for patients who had undergone radiosurgery or surgical resection and are planning adjuvant radiotherapy do not have to have visible disease.
* Patients must have a gadolinium contrast-enhanced three-dimensional MRI scan, whether diagnostic or a MR simulation scan
* Karnofsky performance status of >= 70 or ECOG >= 2
* Patients may have had prior therapy for brain metastasis, including radiosurgery, as long as with hippocampal-sparing, and surgical resection; patients must have completed prior therapy (no specific time lapse between prior treatment and this treatment)

Exclusion Criteria:

* Prior external beam radiation therapy to the brain or whole brain radiation therapy, unless radiosurgery with hippocampal-sparing
* Radiographic evidence of hydrocephalus or other architectural distortion of the ventricular system, including placement of external ventricular drain or ventriculoperitoneal shunt
* Patients with definitive leptomeningeal metastases
* Contraindication to magnetic resonance (MR) imaging such as implanted metal devices or foreign bodies
* Contraindication to gadolinium contrast administration during MR imaging, such as allergy or insufficient renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to Neurocognitive Failure | Baseline, 3 months, 6 months, 12 months (+/- 2 weeks)
  Neurocognitive failure is defined as the first failure, defined as a neurocognitive decline in at least one of the following tests; Hopkins Verbal Learning Test for total recall, delayed recall and delayed recognition; Controlled oral word association; Trail making tests part A and B; Brief visuospatial memory test revised.

SECONDARY OUTCOMES:
Rate of Neurocognitive Preservation | Baseline, 3 months, 6 months, 12 months (+/- 2 weeks)
  Neurocognitive failure is defined as the first failure, defined as a neurocognitive decline in at least one of the following tests; Hopkins Verbal Learning Test for total recall, delayed recall and delayed recognition; Controlled oral word association; Trail making tests part A and B; Brief visuospatial memory test revised.
Change from M.D. Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom Severity Score | Baseline, 3 months, 6 months, 12 months (+/- 2 weeks)
  M.D. Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom Severity Score is a 28-item multi-symptom patient-reported outcome that measures severity of symptoms experience by patients, 9 specific items for patients with brain tumors. Each item ranges from 0 (best condition) to 10 (worst condition). A subscale score (Symptom Severity) is the average of the subscale items, given that a specified minimum numbers of items were completed.
Intracranial Progression-Free Survival | Baseline, 3 months, 6 months, 12 months (+/- 2 weeks)
  Intracranial progression-free survival time defined as time from registration to the date of progression in the brain or death from any cause. Overall survival rates are estimated by Kaplan-Meier method. Patients last known to be alive with be censored at date of last contact. Analysis will be planned after neurocognitive failure is reported.
Overall Survival | Baseline, 3 months, 6 months, 12 months (+/- 2 weeks)
  Overall survival time defined as time from registration to the date of death from any cause. Overall survival rates are estimated by Kaplan-Meier method. Patients last known to be alive with be censored at date of last contact. Analysis will be planned after neurocognitive failure is reported.
Number of Patients with Grade3+ Adverse Event | Baseline, 3 months, 6 months, 12 months (+/- 2 weeks)
  Adverse events will be graded using Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to severity of adverse event; graded from 1 to 5. Grade 1 mild, Grade 2 moderate, Grade 3 severe, Grade 4 life-threatening/disabling, Grade 5 death related to adverse event

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual patient data available to other researchers

REFERENCES:
- [Background] Brown PD, Gondi V, Pugh S, Tome WA, Wefel JS, Armstrong TS, Bovi JA, Robinson C, Konski A, Khuntia D, Grosshans D, Benzinger TLS, Bruner D, Gilbert MR, Roberge D, Kundapur V, Devisetty K, Shah S, Usuki K, Anderson BM, Stea B, Yoon H, Li J, Laack NN, Kruser TJ, Chmura SJ, Shi W, Deshmukh S, Mehta MP, Kachnic LA; for NRG Oncology. Hippocampal Avoidance During Whole-Brain Radiotherapy Plus Memantine for Patients With Brain Metastases: Phase III Trial NRG Oncology CC001. J Clin Oncol. 2020 Apr 1;38(10):1019-1029. doi: 10.1200/JCO.19.02767. Epub 2020 Feb 14. PMID 32058845